CLINICAL TRIAL: NCT01600976
Title: A Phase I Study to Assess the Safety and Pharmacokinetics of Telaprevir (VX-950) in Subjects With Moderate and Severe Hepatic Impairment
Brief Title: A Study to Assess Safety and Pharmacokinetics of Telaprevir in Patients With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Infectious Diseases BVBA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100872; VX-950HPC1001 (Other: Janssen Infectious Diseases BVBA); 2012-001627-13 (EudraCT Number)
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Hepatic Impairment
Keywords: Hepatic impairment; Hepatitis C; Telaprevir; VX-950; Pharmacokinetics; Safety; Unbound plasma concentrations; Child-Pugh score
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): 10 patients with moderate hepatic impairment (CPB [Child-Pugh score 7 to 9])
  Interventions: Drug: telaprevir
- Group 2 (Experimental): 10 healthy control patients with normal hepatic function. Each healthy control patient is matched to a patient in Group 1 with respect to sex, age (± 5 years) and body mass index (BMI) (± 15%)
  Interventions: Drug: telaprevir
- Group 3 (Experimental): up to 4 patients with severe hepatic impairment (CPC [limited to Child Pugh score 10 to 12])
  Interventions: Drug: telaprevir

INTERVENTIONS:
Drug: telaprevir — Type=exact number, unit=mg, number=375, form=tablet, route=oral. Multiple doses of 2 oral tablets of telaprevir will be administered every 8 hours on Days 1 to 5 and a single dose of 2 oral tablets of telaprevir will be administered in the morning on Day 6.
  Other Names: VX-950

SUMMARY:
The purpose of this study is to determine whether the pharmacokinetic (what the body does to the drug) parameters of telaprevir are altered in patients with moderate hepatic impairment, compared to the pharmacokinetic parameters in patients with normal liver function, and measure the relative unbound plasma concentrations of telaprevir.

DETAILED DESCRIPTION:
This is a Phase I, open-label (all people know the identity of the intervention) study to investigate the single dose and steady state pharmacokinetics of telaprevir in patients with moderate hepatic impairment, and measure the relative unbound plasma concentrations of telaprevir. In addition, a small group of patients with severe hepatic impairment will be included to further characterize the pharmacokinetics of telaprevir as a function of liver disease. In this study 24 patients will be enrolled. Based upon physical examination and laboratory assessments, patients will be scored and classified into hepatic function groups on the basis of the Child-Pugh classification (Classification is based on Child-Pugh score which is used to assess prognosis of chronic hepatic disease). A Child-Pugh score of 7 to 9 is considered Child-Pugh category B (CPB) and indicative of moderate liver function impairment; a Child-Pugh score of 10 or greater is considered Child Pugh category C (CPC), indicative of severe liver impairment. Hepatic function groups will consists of Group 1: 10 patients with moderate hepatic impairment (CPB 7 to 9]); Group 2: 10 healthy control patients with normal hepatic function. Each healthy control patient is matched to a patient in Group 1 with respect to sex, age (+5 years or -5 years) and body mass index (BMI) (+15% or -15%); Group 3: 4 patients with severe hepatic impairment (CPC [limited to Child Pugh score 10 to 12]). Safety and tolerability evaluations including adverse events, clinical laboratory tests, 12-lead electrocardiogram, vital signs and physical examination will be recorded throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

For Group 1:

* Moderate liver function impairment (Child Pugh score of 7 to 9)
* History of hepatic disease, such as hepatitis B, previous hepatitis C, alcoholic liver disease, autoimmune hepatitis, non-alcoholic fatty liver disease, hereditary/metabolic, cryptogenic, other
* Consistent with the disease process of hepatic impairment and associated symptoms

For Group 2:

- Matched to a patient with moderate hepatic impairment with regards to sex, age (± 5 years), and BMI (± 15%) and healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality

For Group 3:

* Severe liver function impairment (limited to Child Pugh score of 10 to 12)
* Hepatic impairment due to different etiologies such as hepatitis B, previous hepatitis C, alcoholic liver disease, autoimmune hepatitis, non-alcoholic fatty liver disease, hereditary/metabolic, cryptogenic, other
* Consistent with the disease process of hepatic impairment and associated symptoms

Exclusion Criteria:

For Group 1 and 3:

* Has acute infectious hepatitis
* Has grade 3 or 4 encephalopathy
* Has grade 3 or 4 creatinine elevation
* Is an active candidate for liver transplantation
* Has had variceal bleeding or spontaneous bacterial peritonitis

For Group 1 only:

- Has a porta-caval shunt or transjugular intrahepatic porto-systemic shunts

For Group 2:

Has acute hepatitis A or hepatitis B or hepatitis C infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Comparing the maximum plasma analyte concentration (Cmax) of telaprevir in patients of Group 2 and Group 1 | Day 1 (-1 hour, predose, 0, 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 9, 12, 15, 18 hours postdose), Day 2 to Day 5 (predose), Day 6 (-1 hour, predose, 0, 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 9, 12, 15, 18 hours postdose), and Day 7 (24 hour)
  The pharmacokinetic parameter Cmax of telaprevir following administration of single and multiple oral doses of telaprevir in patients with moderate hepatic impairment (CPB [Child-Pugh score 7 to 9]) ie, Group 1, as compared to matched healthy patients ie, Group 2
Comparing the area under the plasma concentration-time curve (AUC8h) of telaprevir in patients of Group 2 and Group 1 | Day 1 (-1 hour, predose, 0, 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 9, 12, 15, 18 hours postdose), Day 2 to Day 5 (predose), Day 6 (-1 hour, predose, 0, 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 9, 12, 15, 18 hours postdose), and Day 7 (24 hour)
  The pharmacokinetic parameter AUC8h will be measured from time of administration up to 8 hours post dose of telaprevir following administration of single and multiple oral doses of telaprevir in patients with moderate hepatic impairment (CPB) ie, Group 1, as compared to matched healthy patients ie, Group 2
Comparing the actual sampling time to reach the maximum plasma analyte concentration (tmax) of telaprevir in patients of Group 2 and Group 1 | Day 1 (-1 hour, predose, 0, 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 9, 12, 15, 18 hours postdose), Day 2 to Day 5 (predose), Day 6 (-1 hour, predose, 0, 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 9, 12, 15, 18 hours postdose), and Day 7 (24 hour)
  The pharmacokinetic parameter tmax will be measured following administration of single and multiple oral doses of telaprevir in patients with moderate hepatic impairment (CPB) ie, Group 1, as compared to matched healthy patients ie, Group 2

SECONDARY OUTCOMES:
Number of adverse events in Group 1 patients as a measure of safety | up to Day 6
  Number of adverse events in Group 1 patients as a measure of safety will be assessed following administration of single and multiple oral doses of telaprevir in patients with moderate hepatic impairment (CPB) ie, Group 1
Comparing unbound fractions of telaprevir in patients of Group 1 and Group 2 | up to Day 6
  The unbound fractions of telaprevir after single and multiple doses of telaprevir in patients with moderate hepatic impairment ie, Group 1, as compared to matched healthy patients ie, Group 2
Comparing any relationship between the measures of hepatic function and selected pharmacokinetic parameters of telaprevir in patients of Group 1 and Group 2 | up to Day 6
  To assess any relationship between the measures of hepatic function (ie, Child-Pugh score, albumin, bilirubin, alpha-1 acid glycoprotein, and prothrombin time) and selected pharmacokinetic parameters of telaprevir in patients with moderate hepatic impairment (CPB) ie, Group 1 and healthy patients ie, Group 2

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Infectious Diseases BVBA Clinical Trial, Study Director — Janssen Infectious Diseases BVBA
Locations (2):
- Prague, Czechia
- Kiel, Germany

REFERENCES:
- [Derived] Ouwerkerk-Mahadevan S, Halabi A, Cieslarova B, Aerts I, Witek J, Van Solingen-Ristea R, Luo D. Pharmacokinetics of bound and unbound telaprevir in cirrhotic patients with moderate and severe hepatic impairment. J Clin Pharmacol. 2015 Oct;55(10):1147-56. doi: 10.1002/jcph.545. Epub 2015 Jul 7. PMID 25975934
- See also: A Phase I study to assess the safety and pharmacokinetics of telaprevir (VX-950) in subjects with moderate and severe hepatic impairment — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3540&filename=CR100872_CSR.pdf